CLINICAL TRIAL: NCT05234619
Title: Early Versus Late Deflation of Distal Tourniquet in Intravenous Regional Anesthesia With and Without Ketorolac in Hand & Forearm Surgery
Brief Title: Early Versus Late Deflation of Distal Tourniquet in IVRA With and Without Ketorolac in Hand & Forearm Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sherif Salah Ismail, resident doctor at anesthesiology& intensive care unit and pain managment department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-21-11-01
Record Dates: First submitted 2021-11-14; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Hand Injuries With Intravenous Regional Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group one ( lidocaine or control LE ) Early deflation (Active Comparator): Patients in group one (lidocaine or control group LE = 20): will receive 2% lidocaine 3mg/kg (maximum 200 mg) then distal tourniquet deflation occurs after 20 minutes.
  Interventions: Drug: Group one ( lidocaine or control LE ) Early deflation
- Group two ( lidocaine , ketorolac LKE) Early deflation (Active Comparator): Patients in group two (lidocaine ketorolac LKE = 20): will receive 2% lidocaine 3mg/kg (maximum 200 mg) plus ketorolac 0.5mg/kg (maximum 30mg) then distal tourniquet deflation occurs after 20 minutes.
  Interventions: Drug: Group two ( lidocaine , ketorolac LKE ) Early deflation
- Group three ( lidocaine Or control LL ) Late deflation (Active Comparator): Patients in group three (lidocaine or control group LL = 20): will receive 2% lidocaine 3mg/kg (maximum 200 mg) then distal tourniquet deflation occurs after 40 minutes.
  Interventions: Drug: Group three ( lidocaine or control LL ) Late deflation
- Group four ( lidocaine , ketorolac LKL ) Late deflation (Active Comparator): Patients in group four (lidocaine ketorolac LKL = 20): will receive 2% lidocaine 3mg/kg (maximum 200 mg) plus ketorolac 0.5mg/kg (maximum 30mg) then distal tourniquet deflation occurs after 40 minutes.
  Interventions: Drug: Group four ( lidocaine , ketorolac LKL ) Late deflation

INTERVENTIONS:
Drug: Group one ( lidocaine or control LE ) Early deflation — This will be conducted on 20 trauma patients group one who will be present for both elective and emergency Hand and Forearm surgery After establishing noninvasive arterial blood pressure, ECG, peripheral oxygen saturation monitoring, two venous cannulae will be inserted: one in a vein in the dorsum of operative hand and the other in the opposite hand for crystalloid infusion.
  The opposite arm will be elevated for 2 minutes, and using an Esmarch bandage, the venous capacitance of the arm will be emptied. Then, a double-pneumatic tourniquet will be applied. The proximal tourniquet will be inflated to a pressure of 250 mmHg and circulatory isolation of the arm will be confirmed by inspection, lack of radial pulse and failure of pulse oximetry tracing of ipsilateral index finger then Esmarch bandage will be released then induction of lidocaine for intravenous regional anesthesia ( Bier block ) and Early deflation of distal tourniquet occurs after 20 minutes of IVRA induction
  Other Names: Group one ( xyloxaine or control LE ) Early deflation
  Arms: Group one ( lidocaine or control LE ) Early deflation
Drug: Group two ( lidocaine , ketorolac LKE ) Early deflation — As the first intervention this will be conducted on group two but ketorolac will be combined with lidocaine in intravenous regional anesthesia
  Other Names: Group two ( xylocaine , Toradol LKE ) Early deflation
  Arms: Group two ( lidocaine , ketorolac LKE) Early deflation
Drug: Group three ( lidocaine or control LL ) Late deflation — As the first intervention this will be conducted on group three but late deflation of distal tourniquet in intravenous regional anesthesia after 40 minutes of induction of lidocaine for IVRA .
  Other Names: Group three ( xylocaine or control LL ) Late deflation
  Arms: Group three ( lidocaine Or control LL ) Late deflation
Drug: Group four ( lidocaine , ketorolac LKL ) Late deflation — As the first intervention this will be conducted on group four but late deflation of distal tourniquet in intravenous regional anesthesia after 40 minutes of induction of lidocaine and ketorolac for IVRA .
  Other Names: Group four ( xylocaine , toradol LKL ) Late deflation
  Arms: Group four ( lidocaine , ketorolac LKL ) Late deflation

SUMMARY:
Bier block , or intravenous regional anesthesia (IVRA), is a method of anesthesia for upper extremity surgeries. IVRA was first described by August Bier in 1908, and after a period of latency, it began to gain widespread use after Holmes reemphasized its use in 1963. Bier blocks are technically easy to perform, and the rates for successful anesthesia approach 98%. Furthermore, when compared with brachial plexus blocks for outpatient hand and upper extremity surgery, IVRA may realize lower costs and faster postanesthesia recovery.

Although a reliable source of anesthesia, IVRA has been associated with some disadvantages. Some patients cannot tolerate the tourniquet-mediated arm pain, and there are also reports of neurologic injury and compartment syndrome caused by the tourniquet. Perhaps the most serious complications associated with IVRA relate to the potential systemic toxicity of the local anesthetics used. If the local anesthetic gains access to a patient's systemic circulation, the central nervous system (CNS) and cardiovascular system can be affected. The CNS is usually affected first, with symptoms including dizziness, tinnitus, perioral paresthesia, and seizures. Anesthetic-induced toxicity of the cardiovascular system may manifest as hypotension, bradycardia, arrhythmias, or cardiac arrest.

Historically, the tourniquet used in IVRA is left inflated for a minimum of 20 minutes. Theoretically, this allows time for the local anesthetic to bind to the tissues and, consequently, prevent a large bolus of drug from entering the systemic circulation. However, this tourniquet time appears to be arbitrary, and no safe time interval between anesthetic drug injection and tourniquet deflation has been established.

DETAILED DESCRIPTION:
This is a prospective Cohort , controlled , single-blinded , randomized study will be carried out at the department of Anesthesia of Sohag University hospital .

This study will be conducted on 80 trauma patients who will be present for both elective and emergency Hand and Forearm surgery ..

The patients will be allocated to one of four groups :

Early deflation occurs after 20 minutes of induction of IVRA Late deflation occurs after 40 - 60 minutes of induction of IVRA

* Group one ( lidocaine or control LE ) Early deflation
* Group two ( lidocaine , ketorolac LKE) Early deflation
* Group three ( lidocaine Or control LL ) Late deflation
* Group four ( lidocaine , ketorolac LKL ) Late deflation

After establishing noninvasive arterial blood pressure, ECG, peripheral oxygen saturation monitoring, two venous cannulae will be inserted: one in a vein in the dorsum of operative hand and the other in the opposite hand for crystalloid infusion.

The opposite arm will be elevated for 2 minutes, and using an Esmarch bandage, the venous capacitance of the arm will be emptied. Then, a double-pneumatic tourniquet will be applied. The proximal tourniquet will be inflated to a pressure of 250 mmHg and circulatory isolation of the arm will be confirmed by inspection, lack of radial pulse and failure of pulse oximetry tracing of ipsilateral index finger then Esmarch bandage will be released.

ELIGIBILITY:
Inclusion Criteria:

* A normal healthy patient or A patient with mild systemic disease
* Aged between 20 and 70 years
* Male or female
* Schedueled for hand or forearm surgery

Exclusion Criteria:

* Severe Raynaud's Disease (intermittent arteriolar vasospasm of the distal limbs after cold or emotional stimuli).
* Sickle Cell Disease (IVRA is relatively contraindicated, unless meticulous exsanguination of the limb takes place prior to cuff inflation).
* Crush injury to the limb, IVRA may provoke further tissue damage secondary to hypoxia.
* Patients should be fasting, as there may be a possibility of conversion to a general anaesthetic, alternatively the patient may require sedation in addition to IVRA to improve co-operation.
* Psychic, uncooperative patients.
* Patient refusal.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficiency of intravenous regional anesthesia assessed by visual analogue scale | 6 months
  Assessment of lidocaine as anesthetic in IVRA on 40 participants on the quality of the sensorial and motor block .
Duration of intravenous regional anesthesia | 6 months
  Assessment of lidocaine as anesthetic in IVRA on 40 participants on the duration of the sensorial and motor block .
Efficacy of intravenous regional anesthesia as regard tolerance of tourniquet pain . | 6 months
  Assessment of lidocaine as anesthetic in IVRA on 40 participants as regard tourniquet pain during hand and forearm surgery .

SECONDARY OUTCOMES:
Role of keterolac as adjuvant to lidocaine in intravenous regional anesthesia as intraoperative & postoperative analgesic | 6 months
  Assessment of ketorolac as analgesic to lidocaine for intravenous regional anesthesia ( IVRA ) in 40 participants as regard intraoperative and postoperative analgesa during hand and forearm surgery .

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Elsaeed, Study Director — Head of Anesthesiology & intensive care unit department
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Early versus Late deflation of Distal tourniquet in Intravenous Regional Anesthesia With and without Ketorolac in Hand & Forearm surgery
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: Early versus Late deflation of Distal tourniquet in Intravenous Regional Anesthesia With and without Ketorolac in Hand & Forearm surgery

REFERENCES:
- [Background] Rosen MA. Anesthesiology: bupivacaine toxicity. West J Med. 1986 May;144(5):598-9. No abstract available. PMID 18749978
- [Background] Guay J. Adverse events associated with intravenous regional anesthesia (Bier block): a systematic review of complications. J Clin Anesth. 2009 Dec;21(8):585-94. doi: 10.1016/j.jclinane.2009.01.015. PMID 20122591
- [Background] Zahavi GS, Dannon P. Comparison of anesthetics in electroconvulsive therapy: an effective treatment with the use of propofol, etomidate, and thiopental. Neuropsychiatr Dis Treat. 2014 Feb 20;10:383-9. doi: 10.2147/NDT.S58330. eCollection 2014. PMID 24591833